CLINICAL TRIAL: NCT05077280
Title: A Phase II Study of Concurrent Stereotactic Body Radiotherapy With Relatlimab and Nivolumab in Patients With Metastatic Uveal Melanoma
Brief Title: A Study of Concurrent Stereotactic Body Radiotherapy With Opdualag in Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.072-2
Record Dates: First submitted 2021-10-05; First posted 2021-10-14 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Uveal Melanoma
Keywords: metastatic
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — Radiosurgery; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- one arm (Experimental): see below
  Interventions: Radiation: stereotactic body radiotherapy; Drug: Immunotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — Stereotactic Body radiotherapy will be given to 1-5 target metastases in 3 doses over 8 days or less. Each dose will be 15Gy for a total dose of 45GY
Drug: Immunotherapy — Opdualag (nivolumab 480mg and relatlimab 160mg) will be given every 4 weeks for two years

SUMMARY:
This is a phase 2 trial of concurrent stereotactic radiation therapy (SBRT) with immunotherapy with relatlimab and nivolumab for up to two years. SBRT will be given in three doses of 15Gy each to 1-5 separate metastases. Opdualag (nivolumab 480mg and relatlimab 160mg) will be given every 4 weeks for two years

DETAILED DESCRIPTION:
Metastatic uveal melanoma has no standard therapy, but there is evidence that both radiation therapy and immunotherapy may be helpful and may be synergistic. This is a phase 2 trial of concurrent stereotactic radiation therapy (SBRT) with immunotherapy with Opdualag (nivolumab 480mg and relatlimab 160mg) for up to two years. SBRT will be given in three doses of 15Gy each to 1-5 separate metastases, limiting the total dosage to 700cc's of normal liver to <15Gy. Opdualag (nivolumab 480mg and relatlimab 160mg) will be given every 4 weeks for two years. Objectives are to determine the safety and tolerability, and iRECIST will be used to determine responses.We will treat up to 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* measurable metastatic uveal melanoma.
* No concomitant therapy.
* Prior PD1 or tebendafesp allowed.
* Performance status 0-1.
* No active Hepatitis B.
* No known HIV infection.
* WBC>2000, ANC>1500, Hgb >8.
* Creatinine < 3 x ULN.
* AST & ALT < 2.5 x ULN Bilirubin < 2 x ULN.
* Albumin >2.9

Exclusion Criteria:

* Liver tumor volume > 50%.
* Active CNS metastases.
* Pregnancy.
* Prior therapy with Opdualag or relatlimab
* Certain autoimmune diseases.
* Previous liver embolization or radiation.
* Use of systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability of the therapy | 5 years
  toxicity measured by CTAE graded 3-5 toxicities

SECONDARY OUTCOMES:
Response rate | 5 years
  iRECIST defined response rates

OTHER OUTCOMES:
Progression-free survival | 5 years
  survival without progressive cancer
Overall survival | 5 years
  survival

CONTACTS AND LOCATIONS:
Overall Officials: David R Minor, MD, Study Chair — California Pacific Med Center Research Inst.
Locations (1):
- California Pacific Medical Center Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No